CLINICAL TRIAL: NCT05949827
Title: Evaluation of the Effect on Nursing Care Specialists of a Device With Specific Light Algorithms to Maintain and Restore Circadian Melatonin Rhythmicity in Critically Ill Patients
Brief Title: Healing Light Algorithms for Nurses in the ICU
Acronym: ENGAGE-ICU
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technische Universität Berlin (Other)
Responsible Party: Principal Investigator, Alawi Luetz, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: 3000709
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Critical Care; Phototherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active Comparator: LSA-1: Light Scheduling Algorithm-1 (LSA-1): High circadian effective irradiances + Blue Enriched Light episodes
  Interventions: Device: Dynamic Light Therapy Device, LSA-1
- Active Comparator: LSA-2: Light Scheduling Algorithm-2 (LSA-2): High circadian effective irradiances without Blue Enriched Light episodes.
  Interventions: Device: Dynamic Light Therapy Device, LSA-2
- Active Comparator: LSA-3: Light Scheduling Algorithm-3 (LSA-3): Irradiance levels comparable to conventional hospital lighting (control group).
  Interventions: Device: Dynamic Light Therapy Device, LSA-3

INTERVENTIONS:
Device: Dynamic Light Therapy Device, LSA-1 — Dynamic Light Therapy
  Groups: Active Comparator: LSA-1
Device: Dynamic Light Therapy Device, LSA-2 — Dynamic Light Therapy
  Groups: Active Comparator: LSA-2
Device: Dynamic Light Therapy Device, LSA-3 — Dynamic Light Therapy
  Groups: Active Comparator: LSA-3

SUMMARY:
The purpose of this study is to investigate the impact of a newly installed device administering a Light Scheduling Algorithm with high circadian effective irradiances to mechanically ventilated patients on the perceived stress among nursing care specialists.

The investigators will further evaluate the impact on commitment to the workplace, meaning of work, and empathy.

DETAILED DESCRIPTION:
Circadian disruption affects most ICU patients and has far-reaching effects on organ functioning. One of the main factors driving negative outcomes among ICU patients is the lack of natural light. Light as a photoperiodic signal has a great impact on the regulation of the epiphyseal melatonin secretion and the entrainment of the day-night rhythm. This is investigated in the context of the Project HEaling LIght Algorithms for the ICU Patient (HELIA-ICU) a randomized controlled trial investigating the relationship between the treatment with a highly specialized light ceiling and the rhythmicity of melatonin levels and subsequently the decreased incidence of delirium in critically ill patients. For this, the light ceiling was installed in two patient treatment rooms. The current study (ENGAGE-ICU) investigates, in this context, the effects the installation of the highly specialized light ceiling on perceived stress and organization-related perceptions and attitudes among nursing care specialists working under the light ceiling.

The introduction of new elements to the workspace is assumed to have a twofold impact on nursing care specialists exposed to the light ceiling: on the one hand, the levels of illuminance will have an instrumental function, allowing a correct and efficient performance of tasks to the nursing care specialists, thus contributing to a reduction of their perceived levels of stress. On the other hand, the mere presence of the light ceiling will have a symbolic function, signaling the commitment of the organization toward patient welfare and innovation. This will impact attitudes toward the organization like commitment to the workplace and meaning of work. Furthermore, this symbolic function will likely also impact the feelings of empathy toward the patients among nursing care specialists.

Following their work schedules, nursing care specialists will be anonymously allocated into 4 treatment groups:

1. working the early shift in rooms with an operating light ceiling irradiating LSA-1 (high circadian effective irradiances + blue Light Intervention) or LSA-2 (high circadian effective irradiances without blue light intervention)
2. working the late or night shift in rooms with an operating light ceiling irradiating LSA-1 (high circadian effective irradiances + blue Light Intervention) or LSA-2 (high circadian effective irradiances without blue light intervention)
3. working in rooms with an operating light ceiling irradiating LSA-3 (standard irradiances)
4. working in conventional rooms, in which no light ceiling has been installed (Control Group).

Main Hypothesis:

Nursing care specialists working under increased irradiance lighting may differ in the perceived levels of stress compared with nursing care specialists working under conventional irradiance lighting.

Secondary Hypotheses:

1. Nursing care specialists working under increased irradiance lighting receiving illumination with increased irradiance and phases of Blue-Enriched White light (LSA-1) differ in the perceived levels of stress and report lower perceived stress compared with nursing care specialists working under conventional irradiance lighting (LSA-3).
2. Nursing care specialists working under increased irradiance lighting receiving illumination with increased irradiance without phases of Blue-Enriched White light (LSA-2) differ in the perceived levels of stress and report lower perceived stress compared with nursing care specialists working under conventional irradiance lighting (LSA-3).
3. Nursing care specialists working in rooms with a newly installed light ceiling differ in their self-reported commitment to the workplace compared with nursing care specialists working in rooms in which the light ceiling has not been installed.
4. Nursing care specialists working in rooms with a newly installed light ceiling differ in their self-reported meaning of work compared with nursing care specialists working in rooms in which the light ceiling has not been installed.
5. Nursing care specialists working in rooms with a newly installed light ceiling differ in their self-reported empathy compared with nursing care specialists working in rooms in which the light ceiling has not been installed.

ELIGIBILITY:
Inclusion Criteria:

* All nursing care specialists working in ward 101i

Exclusion Criteria:

* Refusal to participate in the study

Termination criteria:

* Withdrawal from the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nursing care specialists
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | April 2023 - April 2024
  Assessed through the single-item Perkhofer Stress Scale. The higher the score the higher the perceived stress (1 to 10)

SECONDARY OUTCOMES:
Commitment to the Workplace | April 2023 - April 2024
  Assessed through the corresponding 2-item scale in the Copenhagen Psychosocial Questionnaire (COPSOQ). The higher the score the higher the self-reported commitment to the workplace (1 to 100)
Meaning of Work | April 2023 - April 2024
  Assessed through the corresponding 2-item scale in the Copenhagen Psychosocial Questionnaire (COPSOQ). The higher the score the higher the self-reported perceived meaning of work (1 to 100)
Empathy | April 2023 - April 2024
  Assessed through the corresponding 4-item scale of the Interpersonal Reactivity Index. The higher the score the higher the self-reported empathy (0 to 28)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided